CLINICAL TRIAL: NCT06359587
Title: Re-Purposing the Ordering of Routine Laboratory Testing in Hospitalized Medical Patients in British Columbia
Brief Title: Re-Purposing the Ordering of Routine Laboratory Tests in Hospitals in British Columbia
Acronym: RePORT-BC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Providence Health & Services (Other); Vancouver Coastal Health (Other Government); Fraser Health (Other); Interior Health (Industry); Northern Hospital, Australia (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Island Health (Other)
Responsible Party: Principal Investigator, Anshula Ambasta, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: H22-03005
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2024-12

CONDITIONS: Hospital Acquired Condition
MeSH Terms: conditions — Iatrogenic Disease

STUDY DESIGN:
Intervention Model Description: Intervention Arm (Intervention Bundle Implementation):
  This arm involves the time periods where hospital units are actively receiving the intervention bundle, including healthcare provider (HCP) and patient engagement tools.
  Control Arm (No Intervention Bundle Implementation):
  This arm represents the time periods when the hospital units do not receive the intervention bundle. This time period is the control period. Each hospital will contribute to intervention and control period data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Intervention Bundle Implementation) (Experimental): This arm involves the time periods of the hospital units where the LTO bundle, including healthcare provider and patient engagement tools, is actively implemented.
  Interventions: Behavioral: Laboratory test overuse (LTO) Bundle
- Control Arm (No LTO Bundle Implementation) (No Intervention): This arm represents the time period of hospital units where the LTO bundle is not implemented.

INTERVENTIONS:
Behavioral: Laboratory test overuse (LTO) Bundle — Key Components of the LTO Bundle:
  Educational materials, including an online module, clinical decision support tool, provision of lab utilization (Audit and Feedback) reports for healthcare providers.
  Patient engagement tools, such as videos and educational infographics. System level implementation tools adapted to the local context, including EMR-based tools and order set changes, etc.
  Arms: Intervention Arm (Intervention Bundle Implementation)

SUMMARY:
The goal of this stepped-wedge cluster randomized trial is to assess the impact of a laboratory test overuse intervention bundle on laboratory test utilization in 6 health authorities (16 hospitals) in British Columbia. The main question it aims to answer is if the intervention bundle, inclusive of healthcare provider and patient engagement tools, can be effectively implemented for hospitalized medical inpatients in 16 hospitals across BC and reduce laboratory test over-use. Researchers will compare hospital clusters that receive the intervention at different (sequential) time points to see if there are significant changes in the measured outcomes after the intervention.

DETAILED DESCRIPTION:
This study aims to reduce unnecessary laboratory test use in hospitals using a stepped-wedge cluster randomized trial design. Over-use of laboratory testing in hospitals leads to patient discomfort, disruption of sleep patterns, and is associated with hospital-acquired anemia. The specific tests that the investigators focus on are complete blood count, electrolytes, creatinine, urea, international normalized ratio and partial thromboplastin time. After the initial control period, the investigators will begin with a pilot-phase for a feasibility assessment of the intervention tools. The intervention bundle will then be rolled out sequentially, one cluster (each cluster containing 2-3 hospitals) at a time in 12-week implementation steps.

The intervention bundle will contain tools to promote education around appropriate use of laboratory testing in hospitals (using an online module, clinical decision support tool), will share data on laboratory test utilization patterns locally, and include patient engagement materials (infographic and video).

Local champions in hospitals will form multidisciplinary implementation teams to facilitate adaptation and delivery of implementation tools within local context. A pragmatic stepped-wedge design will be used to implement the intervention bundle in 16 hospitals grouped into 8 clusters.

The first 4 weeks of implementation will be a pre-intervention period, trialing and adapting tools to the local context. Readiness assessments and workflow observations will be conducted to understand organizational readiness for implementation. Clusters will enter the intervention period during the latter 8 weeks of the implementation period where intervention tools will be deployed.

Data will be collected for at least 24 weeks post-implementation, evaluating the impact of tools without dedicated personnel support. Access to educational resources will continue, and laboratory utilization reports will be sent.

ELIGIBILITY:
Participants involved in this study include the following groups: patients and healthcare providers (including learners, physicians and allied health staff)

Inclusion Criteria:

* Patients: The study will include all adult general medical patients that are admitted to the selected hospital during the study period under general internal medicine or family medicine (hospitalist) provider groups.
* Attending Physicians: All physicians who provide patient care in the general internal medicine or family medicine (hospitalist) provider groups in selected hospitals
* Learners and allied health staff (Medical Students/Resident physicians/Clinical Assistants/ Nurse Practitioners, etc.): All those who help take care of patients and can order labs during the study period in the under general internal medicine or family medicine (hospitalist) provider groups in selected hospitals The date range for both groups will extend from May 2024 until study completion in October 2026.

Exclusion Criteria:

* Patients: all patients in specialized medical units (e.g., coronary care, dialysis units, bone marrow transplants units etc.), in critical care, pediatric, obstetrical, surgical, and psychiatric units.
* Patients and Health Care Providers (HCPs) who are not in the internal medicine or family medicine groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700000 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-11-16 (Estimated); Study Completion 2026-11-16 (Estimated)

PRIMARY OUTCOMES:
Change in number of target laboratory tests ordered per patient-day with LTO bundle compared to control period without LTO bundle | 3 years
  The change in the number of the six target laboratory tests with the LTO bundle

SECONDARY OUTCOMES:
Change in number of total laboratory tests ordered per patient-day with the LTO bundle | 3 years
  Change in the number of all common laboratory tests ordered during the study with the LTO bundle
Rate of hospital re-admissions and mortality | 3 years
  Rate of hospital re-admission and mortality rates over study period with LTO intervention bundle
Change in costs associated with routine laboratory testing | 3 years
  Change in costs associated with routine laboratory testing

CONTACTS AND LOCATIONS:
Overall Officials: Anshula Ambasta, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - University Hospital of Northern British Columbia, Prince George, British Columbia
  - Mount St. Joseph's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

REFERENCES:
- [Derived] Ambasta A, Holroyd-Leduc JM, Pokharel S, Mathura P, Shih AW, Stelfox HT, Ma I, Harrison M, Manns B, Faris P, Williamson T, Shukalek C, Santana M, Omodon O, McCaughey D, Kassam N, Naugler C. Re-Purposing the Ordering of Routine Laboratory Tests in Hospitalized Medical Patients (RePORT): protocol for a multicenter stepped-wedge cluster randomised trial to evaluate the impact of a multicomponent intervention bundle to reduce laboratory test over-utilization. Implement Sci. 2024 Jul 2;19(1):45. doi: 10.1186/s13012-024-01376-6. PMID 38956637